CLINICAL TRIAL: NCT06097676
Title: A Randomized, Double Blind, Active and Placebo Controlled, 5 Way Crossover Study to Determine the Abuse Potential of Orally Administered Gabapentin Enacarbil Immediate Release Capsules in Healthy, Nondependent Recreational Drug Users With Sedative Experience
Brief Title: An Abuse Potential Study of Orally Administered HORIZANT in Healthy, Non-dependent, Recreational Drug Users
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Arbor Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: AR26.3031.1
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Abuse Potential
MeSH Terms: interventions — Alprazolam; 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): - Single oral dose
  Interventions: Drug: Placebo
- Alprazolam 2 mg (Active Comparator): * Single oral dose
  * Drug: Alprazolam 2 mg capsule
  Interventions: Drug: Alprazolam 2 mg
- GE-IR 200 mg (Experimental): * Single oral dose
  * Drug: GE-IR 200 mg capsule
  Interventions: Drug: Gabapentin Enacarbil Immediate Release (GE-IR) 200 mg
- GE-IR 450 mg (Experimental): * Single oral dose
  * Drug: GE-IR 450 mg capsule
  Interventions: Drug: Gabapentin Enacarbil Immediate Release (GE-IR) 450 mg
- GE-IR 700 mg (Experimental): * Single oral dose
  * Drug: GE-IR 700 mg capsule
  Interventions: Drug: Gabapentin Enacarbil Immediate Release (GE-IR) 700 mg

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Alprazolam 2 mg — Oral dose of alprazolam 2 mg
  Other Names: Xanax
  Arms: Alprazolam 2 mg
Drug: Gabapentin Enacarbil Immediate Release (GE-IR) 200 mg — Oral dose of GE-IR 200 mg
  Other Names: Horizant
  Arms: GE-IR 200 mg
Drug: Gabapentin Enacarbil Immediate Release (GE-IR) 450 mg — Oral dose of GE-IR 450 mg
  Other Names: Horizant
  Arms: GE-IR 450 mg
Drug: Gabapentin Enacarbil Immediate Release (GE-IR) 700 mg — Oral dose of GE-IR 700 mg
  Other Names: Horizant
  Arms: GE-IR 700 mg

SUMMARY:
The purpose of this study is to assess the abuse potential of gabapentin enacarbil in healthy adult, non-dependent, recreational drug users.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the abuse potential of gabapentin enacarbil immediate-release (GE-IR), the active moiety in Horizant in comparison to placebo and an active control with known abuse potential (i.e., alprazolam).

This study will be a randomized, double-blind, active- and placebo-controlled, 5-way crossover study to determine the abuse potential of gabapentin enacarbil immediate release (GE-IR) relative to alprazolam (active control) and placebo, in nondependent, recreational drug users with sedative drug use experience.

This study will consist of 3 phases: screening, qualification, and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF),
2. Stated willingness to comply with all study procedures and availability for the duration of the study,
3. Male or female, between 18 and 55 years of age, inclusive,
4. Current nondependent, recreational drug user who has used sedative drugs for recreational (nontherapeutic) purposes (i.e., for psychoactive effects) at least 10 times in the subject's lifetime and at least once in the 12 weeks before screening,
5. Body mass index (BMI) within 18.0 kg/m^2 to 36.0 kg/m^2, inclusive,
6. If female, meets 1 of the following criteria:

   1. If of childbearing potential agrees to use 1 of the accepted contraceptive regimens from at least 30 days prior to the first study drug administration, during the study, and for at least 30 days after the last dose of the study drug. An acceptable method of contraception includes 1 of the following:

      * Abstinence from heterosexual intercourse,
      * Hormonal contraceptives (birth control pills, injectable/implantable/insertable hormonal birth control products, transdermal patch),
      * Intrauterine device (IUD; with or without hormones), Or
   2. If of childbearing potential agrees to use a double barrier method (e.g., condom and spermicide) during the study and for at least 30 days after the last dose of study drug. Or
   3. If of non-childbearing potential, defined as surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or is in a postmenopausal state (i.e., at least 1 year without menses without an alternative medical condition and confirmed follicle stimulating hormone (FSH) ≥ 40 milli-International unit/mL (mIU/mL) prior to the first study drug administration),
7. If male and engaging in sexual activity that has the risk of pregnancy must agree to use a double barrier method (e.g., condom and spermicide) and agree to not donate sperm during the study and for at least 90 days after the last dose of the study medication, a male who has a pregnant partner shall be excluded,
8. Healthy, as determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs or clinical laboratory (including hematology, clinical chemistry, urinalysis, and serology [screening visit only]) at screening visit and admission, as applicable, in the opinion of an investigator,
9. Negative Coronavirus disease 2019 (Covid-19) test prior to each admission, as applicable.

Exclusion Criteria:

1. History of significant hepatic, renal, cardiovascular, pulmonary, hematologic, neurological, psychiatric, gastrointestinal, endocrine, immunologic, ophthalmologic, or dermatologic disease of any etiology (including infections),
2. Presence or history of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability with the exception that cholecystectomy is permitted at the discretion of an investigator,
3. Presence of any significant respiratory illness or presence or history of chronic respiratory disease (e.g., upper respiratory illness, sleep apnea, emphysema, asthma) at screening (subjects with acute respiratory illness may be rescheduled upon resolution at the discretion of an investigator),
4. Personal or family history (first degree relatives) of allergy, hypersensitivity, or drug rash with eosinophilia and systemic symptoms (DRESS) syndrome to gabapentin enacarbil, gabapentin or any drug product including anti-convulsants (e.g., alprazolam, carbamazepine) or related drugs (e.g., other benzodiazepines) or known excipients of any of the drug products in this study (e.g., lactose),
5. History of sensitivity to or poor tolerance of gabapentin enacarbil, gabapentin, pregabalin, or alprazolam,
6. Female who is lactating at screening,
7. Female who is pregnant according to the pregnancy test at screening or prior to the first study drug administration or planning to become pregnant within 30 days following the last study drug administration,
8. History of substance or alcohol dependence (excluding nicotine and caffeine) within the past 2 years, as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV), and/or subject has been in a drug or alcohol rehabilitation program within the last 2 years,
9. Subjects with positive urine drug screen (UDS) results at screening and admission will be assessed for inclusion at the discretion of an Investigator. If tetrahydrocannabinol (THC) is positive at admission to the Qualification phase and Treatment phase, as applicable, a cannabis intoxication evaluation will be done by an investigator and subjects may be permitted to continue in the study, rescheduled, or discontinued at the discretion of an investigator. Other positive test results should be reviewed to determine if the subject may be rescheduled, in the opinion of the investigator,
10. Is a heavy smoker (>20 cigarettes per day or nicotine-equivalent) and/or is unable to abstain from smoking or unable to abstain from the use of prohibited nicotine-containing products for at least 1 hour before and 6 hours after study drug administration (including e-cigarettes, pipes, cigars, chewing tobacco, nicotine topical patches, nicotine gum, or nicotine lozenges),
11. Regularly consumes excessive amounts of caffeine or xanthines within 30 days prior to screening, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day,
12. History of suicidal ideation within 24 months or suicidal behaviour within 2 years of screening, showing suicidal tendency as per the Columbia Suicide Severity Rating Scale (C-SSRS) administered at screening, or is currently at risk of suicide in the opinion of an investigator,
13. Presence of clinically significant ECG abnormalities at the screening visit, as defined by medical judgment, Note: QT corrected according to Fridericia's formula (QTcF) interval of >450 msec in male subjects or >470 msec in female subjects will be exclusionary. The ECG may be repeated once for confirmatory purposes if the initial value obtained exceeds the limits specified,
14. Has creatinine clearance ≤60 ml/min as calculated by the Cockcroft-Gault equation,
15. Any history of tuberculosis,
16. Positive screening results to human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B virus surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab) tests,
17. Intake of an investigational product (IP) within 30 days or 5 times the half-life (whichever is longer) prior to screening,
18. Use of any prescription drugs (with the exception of hormonal contraceptives or hormone replacement therapy) in the 30 days prior to the first study drug administration, that in the opinion of an investigator would put into question the status of the subject as healthy,
19. Use of over-the-counter (OTC) products (including herbal preparations and supplements) within 7 days prior to the first study drug administration, with the exception of ibuprofen or acetaminophen,
20. Donation of plasma in the 7 days prior to screening,
21. Blood donation (excluding plasma) of approximately 500 mL of blood in the 56 days prior to screening,
22. Is, in the opinion of an investigator or designee, considered unsuitable or unlikely to comply with the study protocol for any reason,
23. Poor venous access at screening, as judged by an investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences Clinical Kansas, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ABECD: Period 1: Placebo Period 2: Alprazolam 2 mg Period 3: GE-IR 700 mg Period 4: GE-IR 200 mg Period 5: GE-IR 450 mg
- AEBDC: Period 1: Placebo Period 2: GE-IR 700 mg Period 3: Alprazolam 2 mg Period 4: GE-IR 450 mg Period 5: GE-IR 200 mg
- BACED: Period 1: Alprazolam 2 mg Period 2: Placebo Period 3: GE-IR 200 mg Period 4: GE-IR 700 mg Period 5: GE-IR 450 mg
- BCADE: Period 1: Alprazolam 2 mg Period 2: GE-IR 200 mg Period 3: Placebo Period 4: GE-IR 450 mg Period 5: GE-IR 700 mg
- CBDAE: Period 1: GE-IR 200 mg Period 2: Alprazolam 2 mg Period 3: GE-IR 450 mg Period 4: Placebo Period 5: GE-IR 700 mg
- CDBEA: Period 1: GE-IR 200 mg Period 2: GE-IR 450 mg Period 3: Alprazolam 2 mg Period 4: GE-IR 700 mg Period 5: Placebo
- DCEBA: Period 1: GE-IR 450 mg Period 2: GE-IR 200 mg Period 3: GE-IR 700 mg Period 4: Alprazolam 2 mg Period 5: Placebo
- DECAB: Period 1: GE-IR 450 mg Period 2: GE-IR 700 mg Period 3: GE-IR 200 mg Period 4: Placebo Period 5: Alprazolam 2 mg
- EADBC: Period 1: GE-IR 700 mg Period 2: Placebo Period 3: GE-IR 450 mg Period 4: Alprazolam 2 mg Period 5: GE-IR 200 mg
- EDACB: Period 1: GE-IR 700 mg Period 2: GE-IR 450 mg Period 3: Placebo Period 4: GE-IR 200 mg Period 5: Alprazolam 2 mg
Period: Overall Study
Arm/Group | ABECD | AEBDC | BACED | BCADE | CBDAE | CDBEA | DCEBA | DECAB | EADBC | EDACB
Started | 6 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5
Completed | 6 | 5 | 5 | 5 | 5 | 4 | 5 | 4 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects in the treatment phase (randomized population)
Groups:
- Treatment Phase: Subjects randomized in the treatment phase
Arm/Group | Treatment Phase
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (6.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 40
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Sedative Drug Use In the Past 12 Weeks [Median (Full Range); unit: times] | 12 [1 to 60]

OUTCOME MEASURES:

1. Primary Outcome: Drug Liking "at This Moment" Visual Analog Scale (VAS)
Description: Mean difference in Drug Liking Emax over 24 hours for Drug Liking ("At this moment, my liking for this drug is"), assessed on a bipolar (0 to 100 points; 0: Strong disliking, 50: Neither like nor dislike, 100: Strong liking) VAS.
Time Frame: approximately 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, and 24 hours postdose in the treatment phase and per period of the treatment phase
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Alprazolam 2 mg | GE-IR 200 mg | GE-IR 450 mg | GE-IR 700 mg
Number analyzed (Participants) | 47 | 47 | 47 | 47 | 47
score on a scale | 54.1 (1.47) | 83.8 (1.93) | 58.9 (1.93) | 58.4 (1.5) | 68.5 (2.62)

2. Secondary Outcome: Overall Drug Liking VAS
Description: Mean difference in Emax for Overall Drug Liking ("Overall, my liking for this drug is"), assessed on a bipolar (0 to 100 points; 0: Strong disliking, 50: Neither like nor dislike, 100: Strong liking) VAS.
Time Frame: approximately 12 and 24 hours postdose in the treatment phase and per period of the treatment phase
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Alprazolam 2 mg | GE-IR 200 mg | GE-IR 450 mg | GE-IR 700 mg
Number analyzed (Participants) | 47 | 47 | 47 | 47 | 47
score on a scale | 54.2 (1.71) | 86.6 (2.12) | 62.8 (2.56) | 61.7 (2.4) | 68.2 (3.26)

3. Secondary Outcome: Take Drug Again VAS
Description: Mean difference in Emax for Take Drug Again ("I would take this drug again"), assessed on a bipolar (0 to 100 points; 0: Definitely would not 50: Neither would nor would not, 100: Definitely would) VAS.
Time Frame: approximately 12 and 24 hours postdose in the treatment phase and per period of the treatment phase
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Alprazolam 2 mg | GE-IR 200 mg | GE-IR 450 mg | GE-IR 700 mg
Number analyzed (Participants) | 47 | 47 | 47 | 47 | 47
score on a scale | 55.2 (2.55) | 87.4 (2.14) | 64.6 (2.82) | 65.4 (2.76) | 71.4 (3.52)

4. Secondary Outcome: High VAS
Description: Mean difference in Emax for High ("At this moment, I'm feeling high"), assessed on a unipolar (0 to 100 points; 0: Not at all, 100: Extremely) VAS.
Time Frame: within 1 hour prior to and approximately 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, and 24 hours postdose in the treatment phase and per period of the treatment phase
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Alprazolam 2 mg | GE-IR 200 mg | GE-IR 450 mg | GE-IR 700 mg
Number analyzed (Participants) | 47 | 47 | 47 | 47 | 47
score on a scale | 5.2 (2.61) | 65.5 (4.05) | 11.7 (2.79) | 12.8 (2.91) | 31.6 (4.56)

ADVERSE EVENTS:
Time Frame: The maximum duration of subject participation was approximately 49 days, including screening.
Arm/Group | Placebo | Alprazolam 2 mg | GE-IR 200 mg | GE-IR 450 mg | GE-IR 700 mg
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/50 | 0/49 | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/50 | 0/49 | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 2/49 | 40/50 | 6/49 | 5/51 | 17/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | Alprazolam 2 mg (N=50) | GE-IR 200 mg (N=49) | GE-IR 450 mg (N=51) | GE-IR 700 mg (N=50)
Somnolence (Nervous system disorders) | 0 | 34 (34) | 3 (3) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 3 (3)
Euphoric mood (Psychiatric disorders) | 1 (1) | 15 (15) | 2 (2) | 0 (0) | 5 (5)
Fatigue (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/76/NCT06097676/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT06097676/SAP_001.pdf